CLINICAL TRIAL: NCT01553955
Title: Efficacy of Training in Preparation of Platelet Rich Plasma Using a Standard Centrifuge and Manual Pipetting Methods
Brief Title: Efficacy of Training in Manual Preparation of Platelet Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peterson, Noel, N.D. (Individual)
Responsible Party: Principal Investigator, Noel Peterson, N.D., Principal Investigator, Peterson, Noel, N.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ManualPRP
Record Dates: First submitted 2012-02-07; First posted 2012-03-14 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2012-03

CONDITIONS: Platelet Rich Plasma Production
Keywords: PRP,; Platelet; Manual
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Venipuncture — Blood draw for purposes of training in platelet rich plasma concentration. Trainees will be in pairs and each will draw blood from the other for use in the concentration process.

SUMMARY:
This is a device study in some respects, in that specialized centrifuges are commonly used to make platelet rich plasma, and we are studying the use of standard laboratory equipment to do so. However, it is primarily interventional in that we will evaluate the percentage success of trainees in the concentration of viable platelets to more than 4X baseline using a generic speed centrifuge and a single spin method.

ELIGIBILITY:
Inclusion Criteria:

* English speaking medical practitioners(N.D., D.O. or M.D.)or their office staff

Exclusion Criteria:

* History of difficult blood draws
* Platelet count < 150,000

  * Hb < 37%
* History of blood disorder
* History of altered platelet function
* History of chemotherapy or radiation therapy.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Platelet Concentration Ability After 8 Hours of Training. | 8 Hours After Onset of Training
  Evaluate the percentage success of trainees in the concentration of viable platelets to more than 4X baseline using a generic speed centrifuge and a single spin method. The number evaluated to determine success will be the average concentration ratio achieved in three consecutive concentrations.

SECONDARY OUTCOMES:
Retention of Platelet Concentration Ability At One Month. | Minimum 30 days after training day.
  Evaluate the percentage success of trainees in the concentration of viable platelets to more than 4X baseline using a generic speed centrifuge and a single spin method. The number evaluated to determine success will be the average concentration ratio achieved in three consecutive concentrations performed 30 days or longer after the training day.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Peterson, N.D., Principal Investigator — Noel Peterson, N.D.; K. Dean Reeves, M.D., Study Chair — K. Dean Reeves, M.D., P.A.
Locations (1):
- Noel Peterson, N.D., Lake Oswego, Oregon, United States